CLINICAL TRIAL: NCT01038622
Title: Randomized Directed Immuno Nutrition by L-arginine for Critically Ill Patients
Brief Title: Directed Immuno Nutrition by L-arginine for Critically Ill Patients
Acronym: Immunolarg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P090203
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2009-12

CONDITIONS: Critically Ill
Keywords: L-arginine; Nasal NO; Nosocomial infection; Immune function; HLA-DR expression; Critically ill; Medical ICU patients
MeSH Terms: conditions — Critical Illness; Cross Infection | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-arginine (Active Comparator): 5-day L-arginine treatment (200 mg/kg)
  Interventions: Drug: L-arginine
- placebo (Placebo Comparator): 5-day placebo treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: L-arginine — 5-day L-arginine treatment
  Arms: L-arginine
Drug: placebo — 5-day placebo treatment
  Arms: placebo

SUMMARY:
The main objective of this proof-of-concept study is to demonstrate that the only administration of L-arginine, based on a suspected deficit monitored by nasal nitric oxide measurement, can improve immune functions in critically ill patients at high risk of nosocomial infection.

DETAILED DESCRIPTION:
Background : A meta-analysis has demonstrated the beneficial effect of immuno nutrition in surgical patients, leading to half reduction of incidence of nosocomial infections (HEYLAND DK, JAMA ; 2001). This beneficial effect seems to be related to L-arginine content of formula. In medical intensive care, such an improvement has not been shown, in spite of similar impairment of immune response, which could be due to a more heterogenous population. Our hypothesis is that this beneficial effect could be observed in selected patients of medical intensive care units. L-arginine is a semi-essential amino acid that is the precursor of nitric oxide (NO) synthesis. NO is involved in immune response regulation and has antimicrobial properties, notably into airways where it can be measured in exhaled gas. A decrease in exhaled and nasal NO has been demonstrated in critically ill patients, which may suggest an impairment of its production.

Objectives : The aim of this study is to evaluate the immune effects of enteral L-arginine administration in non surgical critically ill patients. These patients will be selected based on the decrease in nasal NO: directed immuno nutrition. The main objective is to demonstrate that L-arginine administration, as compared to placebo administration, increases nasal NO and enhances immune functions (increase in HLA-DR expression on monocytes, modification of circulating Myeloid-Derived Suppressor Cells (MDSC), decrease in IL-6, IL-17 plasmatic concentrations): stimulation of immune response. The secondary objective is to demonstrate the safety of L-arginine administration on organ failure and on the incidence of nosocomial infections.

This is a monocentric therapeutic trial, randomized and double blind: standard enteral nutrition plus L-arginine (200 mg/kg/d for 5 days from the admission in ICU) versus standard enteral nutrition plus placebo.

Methods-Patients: Non surgical patients admitted in a single medical intensive care unit, under mechanical ventilation for an expected duration > 2 days, with decreased concentrations of nasal NO (< 60 ppb), without severe sepsis or septic shock, will be enrolled. On admission (before treatment), the severity will be evaluated (SAPS II and SOFA score) together with an assessment of plasmatic L-arginine, cytokines (IL-6, IL-17), MDSC, and expression of HLA-DR by monocytes. The same evaluation will be repeated on day 4 (during treatment) and on day 7 (after treatment). The enrolment of 50 patients is statistically enough to demonstrate an increased expression of HLA-DR in the L-arginine group as compared to the placebo group on day 4.

Expected results and perspectives: The aim of this study is to demonstrate the validity of the concept of directed immune stimulation by the sole L-arginine in medical intensive care unit, the patients being selected based on their decrease in exhaled and nasal NO concentrations. This pathophysiological study is the necessary first step before conducting a large clinical trial aimed at demonstrating a reduction of nosocomial infection incidence by L-arginine.

ELIGIBILITY:
Inclusion criteria :

* age > 18 years
* medical patient (absence of recent surgery or trauma)
* initial aggression < 5 days
* mechanically ventilated with expected duration of mechanical ventilation > 2 days
* enteral nutrition
* absence of previous immunosuppression
* nasal NO on day 1 of ICU stay < 60 ppb

Exclusion criteria :

* severe sepsis
* septic shock
* condition associated with a decreased nasal NO concentration (cystic fibrosis, nasal polyposis, primary ciliary dyskinesia
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Expression of HLA-DR in the L-arginine group as compared to the placebo group | on day 3

SECONDARY OUTCOMES:
HLA-DR on day 7, IL-10 and IL-17 on day 3 and 7, MDSC on day 3 and 7 | on day 3 and on day 7
Nosocomial infections | in the first 15 days
Safety issue: organ failure score (SOFA score) on day 3 and 7; issue from ICU | on day 3 and 7

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc TADIE, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Medical Intensive Care Unit, Pompidou Hospital, Paris, France

REFERENCES:
- [Result] Marik PE, Zaloga GP. Immunonutrition in critically ill patients: a systematic review and analysis of the literature. Intensive Care Med. 2008 Nov;34(11):1980-90. doi: 10.1007/s00134-008-1213-6. Epub 2008 Jul 15. PMID 18626628
- [Derived] Tadie JM, Cynober L, Peigne V, Caumont-Prim A, Neveux N, Gey A, Guerot E, Diehl JL, Fagon JY, Tartour E, Delclaux C. Arginine administration to critically ill patients with a low nitric oxide fraction in the airways: a pilot study. Intensive Care Med. 2013 Sep;39(9):1663-5. doi: 10.1007/s00134-013-2984-y. Epub 2013 Jun 19. No abstract available. PMID 23778831